CLINICAL TRIAL: NCT06619444
Title: Dose-Response to Resistance Exercise on Cardiovascular Health
Acronym: DoReps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of California, Riverside (Other); Iowa State University (Other); Harvard School of Public Health (HSPH) (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Duck-chul Lee, Director of Physical Activity Research Center, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24070155; R01HL171098 (NIH)
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Risk
Keywords: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Aerobic Exercise (AE) only (Experimental): Aerobic exercise (AE) training will consist of 60 min of treadmill, elliptical, or bike exercise at a moderate to vigorous (50-80% of heart rate reserve). Intensity of the exercise sessions will be built of gradually. Sessions will occur 2 times per week for the duration of the year.
  Interventions: Behavioral: Aerobic exercise only
- 30 min of resistance exercise (RE) (Experimental): 30 min of resistance exercise (RE) will consist of 30 total minutes of resistance exercise each week (15 min each session) in addition to 60 min of aerobic exercise (AE) each week (30 min each session). Each 15 min session of RE will consist of 2 sets of 8-15 repetitions at 50-80% of 1-rep max of 4 exercises. AE will consist of treadmill, elliptical, or bike exercise at moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be increased gradually. With 1 min rest between sets, this plan is estimated to take approximately 45 min per session. Sessions will occur 2 times per week for the duration of 1 year.
  Interventions: Behavioral: 30 min of resistance exercise
- 60 min of resistance exercise (RE) (Experimental): 60 min of resistance exercise (RE) will consist of 60 total minutes of resistance exercise each week (30 min each session) in addition to 60 min of aerobic exercise each week (30 min each session). Each 30 min session of resistance exercise will consist of 2 sets of 8-15 repetitions at 50-80% of 1-rep max of 8 exercises. Aerobic exercise will consist of treadmill, elliptical, or bike exercise at moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be increased gradually. With 1 min rest between sets, this plan is estimated to take approximately 60 min per session. Sessions will occur 2 times per week for the duration of 1 year.
  Interventions: Behavioral: 60 min of resistance exercise
- 120 min of resistance exercise (RE) (Experimental): 120 min of resistance exercise (RE) will consist of 120 total minutes of resistance exercise each week (60 min each session) in addition to 60 min of aerobic exercise each week (30 min each session). Each 60 min session of resistance exercise will consist of 3 sets of 8-15 repetitions at 50-80% of 1-rep max of 10 exercises. Aerobic exercise will consist of treadmill, elliptical, or bike exercise at moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be increased gradually. With 1 min rest between sets, this plan is estimated to take approximately 90 min per session. Sessions will occur 2 times per week for the duration of 1 year.
  Interventions: Behavioral: 120 min of resistance exercise

INTERVENTIONS:
Behavioral: Aerobic exercise only — Aerobic exercise training will consist of 60 min of treadmill, elliptical, or bike exercise at a moderate to vigorous (50-80% of heart rate reserve). Intensity of the exercise sessions will be built of gradually. Sessions will occur 2 times per week for the duration of the year trial
  Other Names: Aerobic Exercise
  Arms: Aerobic Exercise (AE) only
Behavioral: 30 min of resistance exercise — 30 min of resistance exercise (RE) will consist of 30 total minutes of resistance exercise each week (15 min each session) in addition to 60 min of aerobic exercise each week (30 min each session). Each 15 min session of resistance exercise will consist of 2 sets of 8-15 repetitions at 50-80% of 1-rep max of 4 exercises. Aerobic exercise will consist of treadmill, elliptical, or bike exercise at moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be increased gradually. With 1 min rest between sets, this plan is estimated to take approximately 45 min per session. Sessions will occur 2 times per week for the duration of 1 year.
  Other Names: resistance training
  Arms: 30 min of resistance exercise (RE)
Behavioral: 60 min of resistance exercise — 60 min of resistance exercise (RE) will consist of 60 total minutes of resistance exercise each week (30 min each session) in addition to 60 min of aerobic exercise each week (30 min each session). Each 30 min session of resistance exercise will consist of 2 sets of 8-15 repetitions at 50-80% of 1-rep max of 8 exercises. Aerobic exercise will consist of treadmill, elliptical, or bike exercise at moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be increased gradually. With 1 min rest between sets, this plan is estimated to take approximately 60 min per session. Sessions will occur 2 times per week for the duration of 1 year.
  Other Names: resistance training
  Arms: 60 min of resistance exercise (RE)
Behavioral: 120 min of resistance exercise — 120 min of resistance exercise (RE) will consist of 120 total minutes of resistance exercise each week (60 min each session) in addition to 60 min of aerobic exercise each week (30 min each session). Each 60 min session of resistance exercise will consist of 3 sets of 8-15 repetitions at 50-80% of 1-rep max of 10 exercises. Aerobic exercise will consist of treadmill, elliptical, or bike exercise at moderate to vigorous intensity (50-80% of heart rate reserve). Intensity of the exercise sessions will be increased gradually. With 1 min rest between sets, this plan is estimated to take approximately 90 min per session. Sessions will occur 2 times per week for the duration of 1 year.
  Other Names: resistance training
  Arms: 120 min of resistance exercise (RE)

SUMMARY:
A large body of evidence indicates numerous health benefits of physical activity, including prevention of cardiovascular disease (CVD), the leading cause of death in the US. This evidence has led to US Physical Activity Guidelines that recommend ≥150 min/week of moderate or ≥75 min/week of vigorous aerobic exercise (AE), plus resistance exercise (RE; such as weight lifting) on ≥2 days/week. To date, current research has mostly focused on AE, and we know a great deal about the dose-response relation between AE and health, resulting in clear and practical guidance to the public on the recommended "dose" in min/week. However, currently far less is known about the dose-response for RE: ≥2 days/week are recommended, but with no duration specified. Thus, this project aims to provide clarity on the dose relationship between RE and health. This project will significantly contribute to developing more effective CVD prevention approaches, advancing prescriptive intervention guidelines, by helping to fill the important gaps in knowledge on effective minimum dose, beneficial optimal dose, and safe maximum dose of RE for CVD prevention. Thus, advancing prescriptive intervention guidelines, and provide important insights for future science of physical activity and health.

DETAILED DESCRIPTION:
Participants will be randomly assigned to 1 of four research conditions at varying dosage of resistance exercise (RE) for the duration of 1 year, either 0 min, 30 min, 60 min or 120 min of weekly RE in addition to 60 min of weekly aerobic exercise (AE). Total exercise duration will be split between 2 weekly sessions. Participants in all four groups will receive healthy lifestyle education sessions, and will track daily steps, food intake and activity levels throughout the 1-year intervention. Participants will also complete baseline, 6-month, and 12-month physical examinations, which will include assessments of blood pressure, blood lipids, body composition, and aerobic and muscular fitness. During the first 6 months of intervention will occur in a supervised lab-based setting. Changes in Cardiovascular disease (CVD) risk factors, as well as potential mechanisms (arterial stiffness and inflammatory markers) that might explain a J-shaped dose-response, from baseline to 6 months will be assessed in each of the 4 groups. The second 6 months will follow the same exercise intervention as the first 6 months. However, all participants will be provided with a free health club membership. The second 6 months will be used to investigate the RE dose associated with best adherence in a free-living environment during the second 6 months. In addition, all measures taken at 6 months will also be assessed again at 12 months to examine the long-term effects of different doses of RE as secondary outcomes, given that compliance will not be tightly "enforced" by staff in this unsupervised free-living condition. In this case, the investigators will further carefully consider exercise adherence in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Non-Smoker
* Overweight or Obese: Body Mass Index 25-43 kg/m2
* Inactive: not meeting the US resistance and aerobic exercise guidelines over the last 6 months
* Walking <7,000 steps/day at baseline
* Capable of performing the required exercise training

Exclusion Criteria:

Absolute

* Unstable coronary heart disease or heart failure
* Uncontrolled arrhythmias or severe aortic stenosis
* Acute myocarditis, endocarditis, or pericarditis
* Cancer, requiring treatment in the past 5 years
* Autoimmune diseases, affecting immune system
* Plans to be away ≥4 weeks in the next 1 year
* Pregnancy/anticipated pregnancy during the study
* Other medical condition that is life-threatening or can interfere with or be aggravated by the exercise training
* Uncontrolled Diabetes (HbA1c ≥8.0),
* Hypertensive Blood Pressure ≥160 mm Hg Systolic and/or 100 mm Hg Diastolic,

Relative (should consult a physician)

* Major risk factors for coronary heart disease
* Uncontrolled diabetes or musculoskeletal limitations

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in composite cardiovascular risk score at 6 months | Baseline and 6 months
  The primary outcome will be change from baseline to 6 months in the average composite cardiovascular disease (CVD) risk z-score comprising systolic Blood pressure (SBP), Low-Density lipoprotein cholesterol (LDL-C), fasting glucose, and percent body fat; lower scores indicate better overall CVD risk profile. Each CVD risk factor at baseline and 6 months will be individually standardized to sex-specific z -scores with a mean of 0 and standard deviation (SD) of 1 based on the formula (observed value-mean)/SD for each participant, using the baseline means and SDs from the entire sample.

SECONDARY OUTCOMES:
Change from baseline in arterial stiffness at 6 months | Baseline and 6 months
  Primary outcome will assess changes in all 4 groups from baseline to 6 months on aortic arterial stiffness (purse wave velocity).
Change from baseline in inflammatory markers at 6 months | Baseline and 6 months
  Outcome will assess changes in all 4 groups from baseline to 6 months inflammatory markers (e.g., C-reactive protein, Interleukin 6, Tumor Necrosis Factor alpha).

OTHER OUTCOMES:
Adherence to resistance exercise associated with dose prescription at 12 months | 6 months and 12 months
  This secondary outcome seeks to assess the resistance exercise dose associated with the best adherence to the resistance exercise training prescription during the self-maintenance period of months 6 to 12.

CONTACTS AND LOCATIONS:
Overall Officials: Duck-chul Lee, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Physical Activity Research Center (PARC), Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Datasets will be available to outside researchers and public health professionals through the web sites of the ClinicalTrials.gov and The Physical Activity Research Center (PARC) at the University of Pittsburgh. Outside researchers can learn what data are available and request a de-identified dataset (stripped of all personal health identifiers). All outside investigators must pass an NIH-approved equivalent course on the Protection of Human Subjects. All data requests will be discussed with the research team and approval will be obtained from the institutional review board overseeing the proposal of the data analysis project. Findings from the proposed study will also be disseminated at national and international meetings and publish the findings in peer-reviewed journals. The investigators seek to maximize the knowledge discovered from this study by sharing data to expedite the translation of research into practice to improve cardiovascular health.
Supporting Information: ICF